CLINICAL TRIAL: NCT04741841
Title: Effect of Probiotic Food Supplement "GutMagnific™" in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS), Also Known as Post-viral Fatigue Syndrome, and Comorbid Gastrointestinal Complications
Brief Title: Effect of Probiotics in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImmuneBiotech Medical Sweden AB (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GM_ME/CFS_2020SE
Record Dates: First submitted 2021-01-19; First posted 2021-02-05 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; ME/CFS; Post Viral Fatigue; Post Viral Fatigue Syndrome; Fatigue; Post Exertional Malaise; PEM; Irritable Bowel Syndrome; IBS; Lactobacillus; Probiotic; GutMagnific
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pre-masked randomized vegan capsules with probiotic "GutMagnific" in 2 different doses, or corresponding placebo
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo product is identical to active product in taste and appearance but without probiotic
  Interventions: Dietary Supplement: Placebo
- Treatment high dose (Active Comparator): High dose GutMagnific™
  Interventions: Dietary Supplement: GutMagnific™ H.
- Treatment low dose (Active Comparator): Low dose GutMagnific™
  Interventions: Dietary Supplement: GutMagnific™ L.

INTERVENTIONS:
Dietary Supplement: GutMagnific™ H. — Vegan Capsules with active product, GutMagnific™ high dose
  Arms: Treatment high dose
Dietary Supplement: GutMagnific™ L. — Vegan Capsules with active product, GutMagnific™ low dose
  Arms: Treatment low dose
Dietary Supplement: Placebo — Vegan capsules identical to active product in taste and appearance but without probiotic
  Arms: Placebo

SUMMARY:
Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) is a neurological disease. Currently there is no effective treatment for ME/CFS due to unclear etiology of the disease. The aim of this randomized double-blind placebo-control clinical trial is to study the efficacy of the probiotic food supplement "GutMagnific™" in ME/CFS and comorbid gastrointestinal complications. The outcome of the study will be assessed based on the data from different self-reporting questionnaires and intestinal microbial flora analysis.

DETAILED DESCRIPTION:
Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) is a neurological disease with different symptoms such as fatigue. Symptoms get worse by physical or mental exertion which usually persists for more than 24 hours (post-exertional malaise, PEM). ME/CFS is often characterized by reduced functional capacity, worsening social relationships and reduced ability to cope with work or study.

The exact cause of the ME/CFS is presently unknown however a history of viral infection is common among ME/CFS patients. Prolonged post viral fatigue can develop into a chronic illness and ME/CFS. Current research strongly suggests involvement of gastrointestinal tract and gut microflora disturbances in the pathogenesis with strong evidence supporting the role of imbalance of gut microflora, damaged gut barrier functions and dysfunctional immune responses. There are some features shared with gastrointestinal conditions like irritable bowel syndrome (IBS). GutMagnific™ is an evidence-based probiotic food supplement, scientifically designed to be effective in correcting imbalances of the gut microflora, repairing a damaged gut barrier and reducing inflammation. The strain combination in GutMagnific™ has been carefully designed for its efficacy in IBS and therefore it can be reasonably expected to be also effective in ME/CFS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) at Stora Sköndals Neurological Rehabilitation Clinic
* Gastrointestinal complications similar to IBS

Exclusion Criteria:

* Consumption of any probiotics two weeks before enrolment
* Consumption of other probiotic products during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in ME/CFS symptoms | At the baseline and weekly for 4 months
  ME/CFS symptom rating scale filled up weekly by participants, graded 0-4 to evaluate degree of disease burden, according to the diagnostic Canadian Criteria. Higher score indicating worse outcome.

SECONDARY OUTCOMES:
Changes in Irritable Bowel Syndrome (IBS) symptoms | At the baseline and weekly for 4 months
  Questionnaire for IBS filled up by participants, graded 1-10 to evaluate degree of different bowel symptoms. Higher score indicating better condition.
Changes in the gastrointestinal symptoms based on Rome III criteria | At the baseline and after 3 & 4 months
  Rome III questionnaire for IBS filled up by participants
Changes in health related quality of life (RAND 36-Item Health Survey) | At the baseline and monthly for 4 months
  RAND-36 questionnaire for health-related quality of life filled up by participants. The questionnaire evaluating eight health concepts: physical functioning, role limitations caused by physical health problem, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Possible score is 0 (lowest) to 100 (highest) for each item.
Changes in Hospital Anxiety and Depression Scale (HADS) | At the baseline and after 3 & 4 months
  HADS questionnaire for anxiety and depression filled up by participants.The questionnaire comprises questions for anxiety and depression. Each item on the questionnaire is scored from 0-3 and means that a person can score between 0 and 21 for either anxiety or depression. Higher score representing worse outcome.
Changes in gut microbiota composition | At the baseline and after 3 months
  Fecal samples will be analysed using sequencing-based methods to monitor possible changes related to probiotic treatment. Samples taken prior to and after probiotic treatment in the same participant will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Per Julin, MD/PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Neurological Rehabilitation Clinic in Stora Sköndal, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No